CLINICAL TRIAL: NCT06281652
Title: Cognitive Intervention With Go and Chess in Early and Subjective Cognitive Decline
Acronym: Cognichess
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Cognichess
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Subjective Cognitive Decline
Keywords: Subjective Cognitive Decline; Mild Cognitive Impairment; Cognitive enhancement; Board games
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Go classes (Experimental): Subjects randomized to a group intervention with Go lessons once a week for 12 weeks
  Interventions: Other: Go classes
- Chess classes (Experimental): Subjects randomized to a group intervention with Chess lessons once a week for 12 weeks
  Interventions: Other: Chess classes
- Go & Chess classes (Experimental): Subjects randomized to a group intervention with Go and Chess lessons twice a week for 12 weeks
  Interventions: Other: Go classes; Other: Chess classes
- Control (No Intervention): Subjects randomized to no intervention for 12 weeks

INTERVENTIONS:
Other: Go classes — Classes of board games (Go), performed in groups of 6-10 subjects, once a week
  Arms: Go & Chess classes; Go classes
Other: Chess classes — Classes of board games (Chess), performed in groups of 6-10 subjects, once a week
  Arms: Chess classes; Go & Chess classes

SUMMARY:
The goal of this clinical trial]is to evaluate if learning to play traditional board games could improve cognition in subjects with mild cognitive impairment and subjective cognitive decline. The main questions it aims to answer are:

* Do Go and Chess improve cognition?
* Is a game better than the other? Is the effect of both games on cognition synergistic?
* Do Go and Chess improve quality of life?
* Do Go and Chess improve mood?
* Do Go and Chess improve lifestyle?

Participants will be randomized to one of four groups:

* Group intervention with Go, once a week, for 12 weeks
* Group intervention with Chess, once a week, for 12 weeks
* Group intervention with Go and Chess, twice a week, for 12 weeks
* Control group

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild cognitive impairment or subjective cognitive decline
* Willingness to participate in the board games classes
* Living within 20-minute driving distance from the center
* Signed informed consent

Exclusion Criteria:

* Prior knowledge of the the game rules (in case the subject knows one of the two, they can be randomized to the other one)
* Significant linguistic or sensory impairment (according to clinical judgment)
* Significant behavioral or psychiatric disturbances (according to clinical judgment)
* Significant medical comorbidities (according to clinical judgment)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-02-13 (Estimated); Study Completion 2025-02-13 (Estimated)

PRIMARY OUTCOMES:
General cognition | 12 weeks
  Differences in Montreal Cognitive Assessment between groups [continuous scale, 0-30, higher scores indicate better performances]

SECONDARY OUTCOMES:
Digit Span Forward | 12 weeks
  Differences in Digit Span Forward between groups [continuous scale, 0-9, higher scores indicate better performances]
Digit Span Backwards | 12 weeks
  Differences in Digit Span Backwards between groups [continuous scale, 0-9, higher scores indicate better performances]
Trail Making Test - part A | 12 weeks
  Differences in Trail Making Test - part A between groups [time to complete the task, min 0 seconds, max N/A, higher scores indicate worse performances]
Trail Making Test - part B | 12 weeks
  Differences in Trail Making Test - part B between groups [time to complete the task, min 0 seconds, max N/A, higher scores indicate worse performances]
Semantic fluency | 12 weeks
  Differences in Semantic fluency between groups [continuous scale, min 0, max N/A, higher scores indicate better performances]
Quality of life indicator | 12 weeks
  Differences in WHO Quality of life (WHO-QoL) scale between groups [continuous scale, min 0 max 100, higher scores indicate better quality of life]
Depression | 12 weeks
  Differences in geriatric depression scale scale between groups [continuous scale, min 0 max 15, higher scores indicate worse depression]
Lifestyle | 12 weeks
  Differences in simple lifestyle indicator questionnaire scale between groups [continuous scale, min 0 max 10, higher scores indicate healthier lifestyle]

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Tremolizzo, MD, PhD, Principal Investigator — Fondazione IRCCS San Gerardo
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pozzi FE, Spanio A, Gallo F, Isgro G, Remoli G, Magi A, Moscatelli E, Crisci E, Negro G, Appollonio I, Ferrarese C, Tremolizzo L. Cognitive and social intervention with Go and chess in early and subjective cognitive decline: The COGniChESs study results, with an updated meta-analysis. J Alzheimers Dis. 2026 Jan;109(2):747-756. doi: 10.1177/13872877251401481. Epub 2025 Dec 4. PMID 41342683